CLINICAL TRIAL: NCT05864196
Title: A Phase I/Ib, Single Arm Study of Two Fraction Stereotactic Body Radiation Therapy (SBRT) With Dominant Lesion Simultaneous Integrated Boost (SIB) for the Treatment of Low to Intermediate Risk Prostate Cancer
Brief Title: Two Fraction Prostate SBRT With DIL SIB
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-01306
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer,SBRT,Radiation Treatment,CyberKnife; SBRT; Radiation Treatment; CyberKnife
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men with low to intermediate risk prostate cancer (Experimental): Once a patient is deemed eligible, they will be scheduled for treatment with SBRT, which should be completed within 14 days of screening. Follow up will occur 30 days post radiation and every 4 months, post- radiation for the first 2 years. After the first 2 years of follow up, visits will occur every 6 months until year 5.
  Interventions: Radiation: Two-Fraction Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Two-Fraction Stereotactic Body Radiation Therapy (SBRT) — Two-fraction SBRT with an MRI directed, dominant intraprostatic lesion, simultaneous integrated boost (SIB) based on genomic classification in the treatment of localized prostate cancer.

SUMMARY:
Phase I/Ib, single arm trial of Two-Fraction Stereotactic Body Radiation Therapy (SBRT) with an MRI directed, dominant intraprostatic lesion (DIL), simultaneous integrated boost (SIB) based on genomic classification in the treatment of localized prostate cancer. The primary purpose of this study is to determine the feasibility and safety of two fraction SBRT in patients with localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient age greater than or equal 18
* Localized adenocarcinoma of the prostate
* Biopsy-proven diagnosis of prostate adenocarcinoma
* Low to intermediate risk National Comprehensive Cancer Network (NCCN) disease

  * TX-T2c-8th addition staging
  * PSA<20 ng/ml
  * Grade group 3 or less
* Proper rectal space replacement required as determined by the treating radiation oncologist
* Prostate size less than 60cc defined at time of simulation based on MRI
* Patient ability to undergo MRI and documented dominant Prostate Imaging Reporting and Data System (PI-RADS) 3 or higher lesion

  -- Exception is very low risk, low risk, or favorable intermediate risk with a low to intermediate decipher score in which case an SIB is not utilized
* Androgen-deprivation therapy (ADT) is left to the discretion of the treating radiation oncologist
* Agreement to use effective contraceptive methods such as condoms and spermicidal foam, intrauterine device, or for their partner to use prescription birth control pills
* Ability to give informed consent

Exclusion Criteria:

* High risk disease
* Pelvic lymph node involvement
* Prophylactic lymph node irradiation requirement as determined by the treating radiation oncologist
* Evidence of clinical or radiological extracapsular extension or seminal vesicle invasion
* Prior radiation to the pelvis
* Prior malignancies within the last 5 years
* Inability to meet pre-specified 2 fraction DVH constraints
* Prostate size > 60cc as measures at treatment planning MRI
* Active significant inflammatory bowel disease (IBD) or rheumatological disease
* Prior prostate surgeries

  * Previous uro lift
  * Transurethral resection of the prostate (TURP) within 6 months of SBRT
* "Reasonable" urinary, bowel, and erectile function as defined by the pre-treatment EPIC questionnaire (>50 overall summary score for each domain)
* Men of reproductive potential may not participate unless they agree to use an effective contraceptive method

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Number of Grade 2 or Higher Toxicities per CTCAE version 5.0 | Up to year 5 Post-Treatment
  Number of toxicities determined to be Grade 2 or higher based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Nadir Prostate-Specific Antigen (nPSA) Levels | Up to Year 5 Post-Treatment
  nPSA measured in ng/ml.
Change in Expanded Prostate Cancer Index Composite (EPIC) Quality of Life Questionnaire Score | Baseline, Year 5 Post-Treatment
  61-item assessment of quality of life in prostate cancer patients. The total score is the sum of responses and ranges from 0 to 301; higher scores indicate greater quality of life.
Incidence of Phoenix Definition Biomechanical Failure (BCF) | Up to Year 5 Post-Treatment
  BCF classified as a rise by 2 ng/mL or more in nadir PSA (nPSA).
Disease-Free Survival (DFS) | Up to Year 5 Post-Treatment
  The length of time after SBRT treatment that a patient survives without any signs or symptoms of cancer.
Overall Survival (OS) | Up to Year 5 Post-Treatment
  The length of time after SBRT treatment that a patient survives.
Metastasis-Free Survival (MFS) | Up to Year 5 Post-Treatment
  The length of time after SBRT treatment that a patient is still alive and the cancer has not spread to other parts of the body.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lischalk, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYCyberKnife at Perlmutter Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Vianca.santos@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Vianca.santos@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.